CLINICAL TRIAL: NCT02326051
Title: Timing of Initiation of Low Molecular Weight Heparin Administration in Pregnant Women With Antiphospholipid Syndrome
Brief Title: Timing of Initiation of LMWH Administration in Pregnant Women With APS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MIE2
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Miscarriage; Antiphospholipid Syndrome
Keywords: Antiphospholipid syndrome; APS; LMWH
MeSH Terms: conditions — Abortion, Habitual; Antiphospholipid Syndrome | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Enoxaparin initiation (Active Comparator): Women will start Enoxaparin therapy once positive pregnancy test is established
  Interventions: Drug: Enoxaparin
- Later Enoxaparin initiation (Active Comparator): Women will start Enoxaparin therapy after sonographic confirmation of fetal cardiac pulsation
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Women will start Enoxaparin therapy in a dose of 40 mg/day subcutaneously once positive pregnancy test is established and the therapy will continue until termination of pregnancy
  Other Names: Clexan
  Arms: Early Enoxaparin initiation
Drug: Enoxaparin — Women will start Enoxaparin therapy in a dose of 40 mg/day subcutaneously after sonographic confirmation of fetal cardiac pulsation and the therapy will continue until termination of pregnancy
  Other Names: Clexan
  Arms: Later Enoxaparin initiation

SUMMARY:
Evaluation of the effect of altering the timing of initiation of low molecular weight heparin (LMWH) administration on the pregnancy outcomes in women with antiphospholipid syndrome (APS)

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; one will start Enoxaparin therapy once positive pregnancy test is established and the other will start Enoxaparin therapy after sonographic confirmation of fetal cardiac pulsation. In all women, Enoxaparin will be given in a dose of 40 mg/day subcutaneously and the therapy will continue until termination of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with APS diagnosed according to the revised classification criteria for APS in 2006 in Sydney, Australia
* Early pregnancy body weight is 50-90 Kg

Exclusion Criteria:

* Women with systemic lupus erythematosus (SLE)
* Women with active thromboembolic disorders
* Women with history of previous thromboembolic disorders

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | After 12 weeks gestational age
  Number of pregnancies that progressed beyond the critical first trimester (12 weeks gestational age) per number of pregnant women

SECONDARY OUTCOMES:
Fetal loss | From 20 weeks to 42 weeks gestational age
  Unexplained fetal death of morphologically normal fetus after the first trimester
Preterm delivery | From 20 weeks to 34 weeks gestational age
  Delivery of morphologically normal fetus before 34 weeks of gestation due to severe preeclampsia or placental insufficiency
Intrauterine growth restriction (IUGR) | At birth
  Birth weight less than the 10th percentile for gestational age
Congenital fetal malformations | At birth

OTHER OUTCOMES:
Hemorrhagic complications | After 12 weeks gestational age up to birth
Thromboembolic complications | After 12 weeks gestational age up to birth

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Eid, Dr, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Waleed El-refaie, Dr, Study Director — Mansoura University; Ahmed El-Zayadi, Dr, Study Director — Mansoura University; Ahmed Badawy, Prof, Study Chair — Mansoura University
Locations (2):
- Egypt (2):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Undecided